CLINICAL TRIAL: NCT06869408
Title: Observational Study on the Patient's Ability to Use a Digital Platform in Heart Failure
Acronym: CAP-IC
Status: Completed | Type: Observational
Sponsor: Persei Vivarium (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAP-IC
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Caaring; DTx; real-world data; Digital Health; Remote patient monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Heart Failure has a global prevalence of 1 to 3% in the adult population with an incidence of 1 to 20 cases per 1,000 people. Furthermore, HF is often associated with a number of comorbidities (anaemia, arrhythmias, depression, hyperuricemia, coronary heart disease etc.), which greatly deteriorates the patient's quality of life.

Despite the development of specific drugs, HF has a very high mortality rate, and it is the first cause of unscheduled income. An increase of 50% of these incomes is expected in the next 25 years.

In this context, the use of digital tools/platforms that allow remote monitoring of patients and that facilitate telemedicine have shown potential to improve treatment adherence and facilitate continued therapeutic education, improving clinical results with savings in time and associated costs.

This study focuses on studying the ability of heart failure patients with reduced ejection fraction (EF≤40%) to use a digital platform through an application installed on the patient's smartphone.

DETAILED DESCRIPTION:
This is an observational, prospective, single-center study. The protocol and informed consent document have been reviewed and approved by the Ethical Committee and the study will be performed in accordance with the Declaration of Helsinki

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Informed Consent is obtained from the patient
* Patients diagnosed with heart failure with reduced ejection fraction (EF≤40%)
* Patients who extensively use a smartphone.

Exclusion Criteria:

* Patients who will not be able to commit to carrying out the follow-ups or do not have adequate technological skills.
* Patients with inability to give adequately the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with reduced ejection fraction (EF≤40%)from Hospital Universitario Son Llatzer who met the inclusion criteria and sign the informed consent will be included.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Patients' ability to report data through a digital platform: Clinical situation | Day 0, every 3 days up to week 12
  Percentage of patients with at least 80% of the data completed per form: clinical situation.
Patients' ability to report data through a digital platform: Treatment and adherence | Day 0, and weekly up to week 12
  Percentage of patients with at least 80% of the data completed per form: treatment and adherence.
Patients' ability to report data through a digital platform: Quality of Life | Day 0, Week 4 and Week 12
  Percentage of patients with at least 80% of the data completed of the quality life questionnaire WHOQOL (World Health Organization Quality Of Life)
Patients' ability to report data through a digital platform: Mediterranean Diet Adherence | Day 0, Week 4 and Week 12
  Percentage of patients with at least 80% of the data completed by MEDAS (Mediterranean Diet Adherence Screener) questionnaire
Patients' ability to report data through a digital platform: European Heart Failure Self-Care Behaviour Scale | Day 0, Week 4 and Week 12
  Percentage of patients with at least 80% of the data completed by EHFScB (European Heart Failure Self-Care Behaviour Scale) scale
Patients' ability to report data through a digital platform: Liquid Consumption Questionnaire | Day 0, Week 4 and Week 12
  Percentage of patients with at least 80% of the data completed by Liquid Consumption Questionnaire
Patient participation rate | Week 12
  Patient participation rate defined as the ratio between the questionnaries requested and completed
Percentage of patients with at least 80% of data completed. | Week 12
  Percentage of patients with at least 80% of data completed in the application
Percentage of patients with 100% of data completed. | Week 12
  Percentage of patients with 100% of data completed in the application.

SECONDARY OUTCOMES:
Change in the use of health resources | Day 0 and Mothly up to 3 months
  Change in patient´s use of health resources scores at basal monthly and at the end of the study compared to baseline: Number of visits to specialists (e.g. cardiology, primary care, etc.), number of emergency room visits, or number of hospital readmissions.
  The changes will be measured through a specific form created for this purpose.
Changes in the patient's quality of life scale: WHOQOL | Day 0, week 4 and week 12]
  Changes in patient's quality of life scale WHOQOL (World Health Organization Quality of Life) scores at week 4 and at the end of the study compared to baseline. Values: 0-100, a higher score reflects a better health-related quality of life.
Changes in the patient's MEDAS scale: Adherence to Mediterranean Diet | Day 0, week 4 and week 12
  Changes in patient's scale MEDAS (Mediterranean Diet Adherence Screener) scores at week 4 and at the end of the study compared to baseline. Values: 0-14, a higher score reflects a better the adherence to the Mediterranean Diet.
Changes in the patient's in EHFScB: European Heart Failure Self-Care Behaviour Scale | Day 0, week 4 and week 12
  Changes in patient's EHFScB scale (European Heart Failure Self-Care Behaviour scale) scores at week 4 and at the end of the study compared to baseline. Values: 0-100, a higher score reflects a better Self-Care Behaviour in the standardized score.
Changes in the patient's in Liquid Consumption | Day 0, week 4 and week 12
  Changes in patient's Liquid Consumption Questionnaire. The changes will be measured through a specific form created for this purpose
Changes in the patient's: Adherence to treatment | Day 0, Weekly up to Week 12
  Changes in patient's Adherence to treatment measured by patient self-report. The questionnaire ask for treatments taken or forgotten. Changes will be measured through a specific form created for this purpose
Changes in the patient's Clinical Data | Day 0, every 3 days up to Week 12
  Changes in patient's Clinical data (symptoms related to heart failure) measured through a specific form created for this purpose.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Son Llatzer, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No